CLINICAL TRIAL: NCT02614196
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients With Episodic Migraine - the EVOLVE-2 Study
Brief Title: Evaluation of Efficay & Safety of Galcanezumab in the Prevention of Episodic Migraine- the EVOLVE-2 Study
Acronym: EVOLVE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15768; I5Q-MC-CGAH (Other: Eli Lilly and Company); 2015-001882-17 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor is also masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (6):
- Galcanezumab 120mg (Experimental): Galcanezumab 240mg given as loading dose at first dosing visit followed by galcanezumab 120mg once a month for 5 months by subcutaneous (SC) injection.
  Interventions: Drug: Galcanezumab
- Galcanezumab 240mg (Experimental): Galcanezumab 240mg given by SC injection once a month for 6 months.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo given by SC injection once a month for 6 months.
  Interventions: Drug: Placebo
- Galcanezumab 120mg Maximum Extended Enrollment Cohort (Experimental): Galcanezumab 240mg given as loading dose at first dosing visit followed by galcanezumab 120mg once a month for 5 months by subcutaneous (SC) injection.
  Interventions: Drug: Galcanezumab
- Galcanezumab 240mg Maximum Extended Enrollment Cohort (Experimental): Galcanezumab 240mg given by SC injection once a month for 6 months.
  Interventions: Drug: Galcanezumab
- Placebo Maximum Extended Enrollment Cohort (Placebo Comparator): Placebo given by SC injection once a month for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab 120mg; Galcanezumab 120mg Maximum Extended Enrollment Cohort; Galcanezumab 240mg; Galcanezumab 240mg Maximum Extended Enrollment Cohort
Drug: Placebo — Administered SC
  Arms: Placebo; Placebo Maximum Extended Enrollment Cohort

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of the study drug known as galcanezumab in participants with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta version (1.1 or 1.2) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, migraine onset prior to age 50 and MONTHLY frequency of 4-14 MHD.

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to galcanezumab or another Calcitonin Gene-Related Peptide (CGRP) antibody.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to galcanezumab.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 986 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (99):
- United States (49):
  - 21st Century Neurology, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Axiom Research, Apple Valley, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Pacific Research Partners, LLC, Oakland, California
  - Medical Center for Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Meridien Research, Tampa, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - Diamond Headache Clinic, Chicago, Illinois
  - Josephson Wallack Munshower Neurology, Indianapolis, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Novex Clinical Research, New Bedford, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Healthcare Research Network - Hazelwood, Hazelwood, Missouri
  - Nevada Headache Institute, Las Vegas, Nevada
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Regional Clinical Research, Binghamton, New York
  - SPRI Clinical Trials, LLC., Brooklyn, New York
  - High Point Clinical Trials Center, High Point, North Carolina
  - Neurology & Neuroscience Associates, Inc., Akron, Ohio
  - Univ of Cincinnati College of Medicine, Cincinnati, Ohio
  - Urgent Care Specialists, LLC, Columbus, Ohio
  - Urgent Care Specialists, LLC, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Neurology Associates, Springfield, Oregon
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Mountain View Clinical Research, Inc, Greer, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - FutureSearch Trials, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Clinpoint Trial, LLC, Waxahachie, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - Jordan River Family Medicine, South Jordan, Utah
  - Health Research of Hampton Roads Inc, Newport News, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Polyclinic, Seattle, Washington
  - Dean Foundation for Health Research and Education, Middleton, Wisconsin
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kladno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Königstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prien am Chiemsee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Israel (4):
  - Hillel Yaffe, Hadera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramat Gan
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
- Netherlands (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geleen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tilburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- Puerto Rico (2):
  - Cortex, PSC, Las Piedras
  - SomniCare Sleep Institute, San Juan
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hwaseong-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valladolid
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hull
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liverpool
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ailani J, Kuruppu DK, Rettiganti M, Oakes T, Schroeder K, Wietecha L, Port M, Blumenfeld AM. Does "wearing off" of efficacy occur in galcanezumab-treated patients at the end of the monthly treatment cycle? Post hoc analyses of four phase III randomized trials. Headache. 2022 Feb;62(2):198-207. doi: 10.1111/head.14257. Epub 2022 Jan 25. PMID 35076090
- [Derived] Citrome L, Sanchez Del Rio M, Dong Y, Nichols RM, Tockhorn-Heidenreich A, Foster SA, Stauffer VL. Benefit-Risk Assessment of Galcanezumab Versus Placebo for the Treatment of Episodic and Chronic Migraine Using the Metrics of Number Needed to Treat and Number Needed to Harm. Adv Ther. 2021 Aug;38(8):4442-4460. doi: 10.1007/s12325-021-01848-x. Epub 2021 Jul 15. PMID 34264500
- [Derived] Jedynak J, Eross E, Gendolla A, Rettiganti M, Stauffer VL. Shift from high-frequency to low-frequency episodic migraine in patients treated with Galcanezumab: results from two global randomized clinical trials. J Headache Pain. 2021 May 28;22(1):48. doi: 10.1186/s10194-021-01222-w. PMID 34049484
- [Derived] Pozo-Rosich P, Samaan KH, Schwedt TJ, Nicholson RA, Rettiganti M, Pearlman EM. Galcanezumab Provides Consistent Efficacy Throughout the Dosing Interval Among Patients with Episodic and Chronic Migraine: A Post Hoc Analysis. Adv Ther. 2021 Jun;38(6):3154-3165. doi: 10.1007/s12325-021-01708-8. Epub 2021 May 5. PMID 33950375
- [Derived] Ament M, Day K, Stauffer VL, Skljarevski V, Rettiganti M, Pearlman E, Aurora SK. Effect of galcanezumab on severity and symptoms of migraine in phase 3 trials in patients with episodic or chronic migraine. J Headache Pain. 2021 Feb 6;22(1):6. doi: 10.1186/s10194-021-01215-9. PMID 33549036
- [Derived] Kuruppu DK, North JM, Kovacik AJ, Dong Y, Pearlman EM, Hutchinson SL. Onset, Maintenance, and Cessation of Effect of Galcanezumab for Prevention of Migraine: A Narrative Review of Three Randomized Placebo-Controlled Trials. Adv Ther. 2021 Mar;38(3):1614-1626. doi: 10.1007/s12325-021-01632-x. Epub 2021 Feb 5. PMID 33544305
- [Derived] Dodick DW, Doty EG, Aurora SK, Ruff DD, Stauffer VL, Jedynak J, Dong Y, Pearlman EM. Medication overuse in a subgroup analysis of phase 3 placebo-controlled studies of galcanezumab in the prevention of episodic and chronic migraine. Cephalalgia. 2021 Mar;41(3):340-352. doi: 10.1177/0333102420966658. Epub 2020 Nov 3. PMID 33143451
- [Derived] Ailani J, Andrews JS, Rettiganti M, Nicholson RA. Impact of galcanezumab on total pain burden: findings from phase 3 randomized, double-blind, placebo-controlled studies in patients with episodic or chronic migraine (EVOLVE-1, EVOLVE-2, and REGAIN trials). J Headache Pain. 2020 Oct 17;21(1):123. doi: 10.1186/s10194-020-01190-7. PMID 33069214
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Bangs ME, Kudrow D, Wang S, Oakes TM, Terwindt GM, Magis D, Yunes-Medina L, Stauffer VL. Safety and tolerability of monthly galcanezumab injections in patients with migraine: integrated results from migraine clinical studies. BMC Neurol. 2020 Jan 17;20(1):25. doi: 10.1186/s12883-020-1609-7. PMID 31952501
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569
- [Derived] Silberstein SD, Stauffer VL, Day KA, Lipsius S, Wilson MC. Galcanezumab in episodic migraine: subgroup analyses of efficacy by high versus low frequency of migraine headaches in phase 3 studies (EVOLVE-1 & EVOLVE-2). J Headache Pain. 2019 Jun 28;20(1):75. doi: 10.1186/s10194-019-1024-x. PMID 31253091
- [Derived] Stauffer VL, Wang S, Voulgaropoulos M, Skljarevski V, Kovacik A, Aurora SK. Effect of Galcanezumab Following Treatment Cessation in Patients With Migraine: Results From 2 Randomized Phase 3 Trials. Headache. 2019 Jun;59(6):834-847. doi: 10.1111/head.13508. Epub 2019 Apr 3. PMID 30942898
- [Derived] Forderreuther S, Zhang Q, Stauffer VL, Aurora SK, Lainez MJA. Preventive effects of galcanezumab in adult patients with episodic or chronic migraine are persistent: data from the phase 3, randomized, double-blind, placebo-controlled EVOLVE-1, EVOLVE-2, and REGAIN studies. J Headache Pain. 2018 Dec 29;19(1):121. doi: 10.1186/s10194-018-0951-2. PMID 30594122
- [Derived] Nichols R, Doty E, Sacco S, Ruff D, Pearlman E, Aurora SK. Analysis of Initial Nonresponders to Galcanezumab in Patients With Episodic or Chronic Migraine: Results From the EVOLVE-1, EVOLVE-2, and REGAIN Randomized, Double-Blind, Placebo-Controlled Studies. Headache. 2019 Feb;59(2):192-204. doi: 10.1111/head.13443. Epub 2018 Nov 21. PMID 30462830
- [Derived] Skljarevski V, Matharu M, Millen BA, Ossipov MH, Kim BK, Yang JY. Efficacy and safety of galcanezumab for the prevention of episodic migraine: Results of the EVOLVE-2 Phase 3 randomized controlled clinical trial. Cephalalgia. 2018 Jul;38(8):1442-1454. doi: 10.1177/0333102418779543. Epub 2018 May 31. PMID 29848108
- See also: Click here for more information about this study: Evaluation of Galcanezumab in the Prevention of Episodic Migraine- the EVOLVE-2 Study — http://www.lillytrialguide.com/EN-US/studies/headache/cgah

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; Placebo Maximum Extended Enrollment Cohort: Participants received placebo by subcutaneous injection once a month for 6 months during double blind treatment phase. Participants did not receive any intervention during post-treatment follow-up phase.
- Galcanezumab 120mg; Galcanezumab 120mg Maximum Extended Enrollment Cohort: Participants received loading dose of 240mg galcanezumab at 1st dosing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection during double blind treatment phase. Participants did not receive any intervention during post-treatment follow-up phase.
- Galcanezumab 240mg; Galcanezumab 240mg Maximum Extended Enrollment Cohort: Participants received 240mg galcanezumab by subcutaneous injection once a month for 6 months during double blind treatment phase. Participants did not receive any intervention during post-treatment follow-up phase.
Period: Double Blind Treatment Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Placebo Maximum Extended Enrollment Cohort | Galcanezumab 120mg Maximum Extended Enrollment Cohort | Galcanezumab 240mg Maximum Extended Enrollment Cohort
Started | 463 | 233 | 226 | 30 | 15 | 19
Received at Least One Dose of Study Drug | 461 | 231 | 223 | 30 | 14 | 19
Completed | 387 | 203 | 195 | 26 | 14 | 19
Not Completed | 76 | 30 | 31 | 4 | 1 | 0
Not completed — Adverse Event | 8 | 5 | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 7 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 2 | 1 | 0 | 1 | 0
Not completed — Terminated by sponsor | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 39 | 11 | 14 | 4 | 0 | 0
Not completed — Did not receive study drug | 2 | 2 | 3 | 0 | 0 | 0
Period: Post Treatment Follow-up Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Placebo Maximum Extended Enrollment Cohort | Galcanezumab 120mg Maximum Extended Enrollment Cohort | Galcanezumab 240mg Maximum Extended Enrollment Cohort
Started | 410 (Participants who discontinued double blind phase had an option to enter post treatment phase) | 213 (Participants who discontinued double blind phase had an option to enter post treatment phase) | 207 (Participants who discontinued double blind phase had an option to enter post treatment phase) | 25 (Participants who discontinued double blind phase had an option to enter post treatment phase) | 15 (Participants who discontinued double blind phase had an option to enter post treatment phase) | 19 (Participants who discontinued double blind phase had an option to enter post treatment phase)
Completed | 390 | 208 | 199 | 24 | 13 | 19
Not Completed | 20 | 5 | 8 | 1 | 2 | 0
Not completed — Lost to Follow-up | 8 | 3 | 3 | 0 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 10 | 1 | 5 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug for non-ME2 arms & All randomized participants for ME2 arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Placebo Maximum Extended Enrollment Cohort | Galcanezumab 120mg Maximum Extended Enrollment Cohort | Galcanezumab 240mg Maximum Extended Enrollment Cohort | Total
Number analyzed (Participants) | 461 | 231 | 223 | 30 | 15 | 19 | 979
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.33 (11.30) | 40.91 (11.15) | 41.91 (10.77) | 45.37 (10.30) | 39.40 (11.58) | 42.58 (11.13) | 41.95 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 393 | 197 | 191 | 22 | 13 | 14 | 830
  Male | 68 | 34 | 32 | 8 | 2 | 5 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 118 | 58 | 61 | 4 | 2 | 3 | 246
  Not Hispanic or Latino | 318 | 162 | 151 | 21 | 10 | 12 | 674
  Unknown or Not Reported | 25 | 11 | 11 | 5 | 3 | 4 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 8 | 13 | 0 | 0 | 0 | 41
  Asian | 50 | 28 | 24 | 30 | 15 | 19 | 166
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 36 | 11 | 16 | 0 | 0 | 0 | 63
  White | 325 | 166 | 152 | 0 | 0 | 0 | 643
  More than one race | 30 | 18 | 16 | 0 | 0 | 0 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 22 | 12 | 10 | 0 | 0 | 0 | 44
  South Korea | 34 | 17 | 17 | 14 | 7 | 9 | 98
  Netherlands | 24 | 11 | 11 | 0 | 0 | 0 | 46
  United States | 224 | 112 | 110 | 0 | 0 | 0 | 446
  Czechia | 39 | 19 | 19 | 0 | 0 | 0 | 77
  Taiwan | 12 | 7 | 5 | 16 | 8 | 10 | 58
  Mexico | 36 | 18 | 17 | 0 | 0 | 0 | 71
  United Kingdom | 8 | 4 | 3 | 0 | 0 | 0 | 15
  Israel | 11 | 5 | 5 | 0 | 0 | 0 | 21
  Germany | 37 | 19 | 19 | 0 | 0 | 0 | 75
  Spain | 14 | 7 | 7 | 0 | 0 | 0 | 28
Migraine Headache Days (MHD) per month [Mean (Standard Deviation); unit: Days per Month] — Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Days per Month | 9.19 (2.99) | 9.07 (2.87) | 9.06 (2.92) | 9.16 (2.98) | 9.06 (2.86) | 9.01 (2.90) | 9.10 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Migraine Headache : A headache, with or without aura, of ≥30 minutes duration with both of the following required features (A and B):
  A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity; AND B) During headache at least one of the following: Nausea and/or vomiting; Photophobia and phonophobia;
  Overall mean is derived from the average of months 1 to 6 from mixed model repeated measures (MMRM) model. Least Square (LS) mean was calculated using mixed model repeated measures (MMRM) model with treatment, pooled country, month, and treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
  As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups
Measure: Least Squares Mean (Standard Error); unit: Migraine Headache Days per Month
Groups:
- Placebo: Participants received placebo by subcutaneous injection once a month for 6 months.
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
- Galcanezumab 240mg: Participants received 240mg galcanezumab by subcutaneous injection once a month for 6 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 450 | 226 | 220
Migraine Headache Days per Month | -2.28 (0.20) | -4.29 (0.25) | -4.18 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -2.02, 95% CI 2-sided [-2.55 to -1.48], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -1.90, 95% CI 2-sided [-2.44 to -1.36], Standard Error of Mean 0.27

2. Secondary Outcome: Mean Percentage of Participants With Reduction From Baseline ≥50%, ≥75%, and 100% in Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred.
  Mean is derived from the average of months 1 to 6 from generalized linear mixed model repeated measures. Mean percentages of participants were calculated with a generalized linear mixed model repeated measures method with treatment, month and treatment by month, baseline.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of participants
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 450 | 226 | 220
percentage of participants
  ≥50% | 36 (1.7) | 59.3 (2.4) | 56.5 (2.5)
  ≥75% | 17.8 (1.3) | 33.5 (2.3) | 34.3 (2.3)
  100% | 5.7 (0.7) | 11.5 (1.4) | 13.8 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥50%; Test type: Superiority; Odds Ratio (OR) = 2.60, 95% CI 2-sided [2.03 to 3.32]
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥50%; Test type: Superiority; Odds Ratio (OR) = 2.31, 95% CI 2-sided [1.81 to 2.96]
Statistical Analysis 3: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥75%; Test type: Superiority; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.78 to 3.06]
Statistical Analysis 4: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥75%; Test type: Superiority; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.84 to 3.17]
Statistical Analysis 5: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥100%; Test type: Superiority; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.50 to 3.12]
Statistical Analysis 6: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥100%; Test type: Superiority; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.87 to 3.81]

3. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire (MSQ) Version 2.1 Role Function Restrictive Domain
Description: MSQ v2.1 was developed to address physical & emotional limitations of specific concern to individuals with migraine.
  It consists of 14 items that address 3 domains:(1) Role Function-Restrictive (items 1-7);(2) Role Function- Preventive (items 8-11);&(3) Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated.Total raw scores for each domain is the sum of the final item value for all of the items in that domain.After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
  Mean is derived from the average of months 4 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline by month & baseline MHD category as fixed factors.
Time Frame: Baseline, Month 4 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline value.
  As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants received placebo subcutaneously once a month for 6 months.
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab followed by 120mg galcanezumab once a month for 5 months subcutaneously.
- Galcanezumab 240mg: Participants received 240mg galcanezumab subcutaneously once a month for 6 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 443 | 226 | 219
units on a scale | 19.65 (0.92) | 28.47 (1.15) | 27.04 (1.17)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = 8.82, 95% CI 2-sided [6.33 to 11.31], Standard Error of Mean 1.27
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = 7.39, 95% CI 2-sided [4.88 to 9.90], Standard Error of Mean 1.28

4. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Migraine or Headache
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 6 from MMRM model.LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed effects.
Time Frame: Baseline, Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline value.
  As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Least Squares Mean (Standard Error); unit: Days per Month
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months subcutaneously.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 450 | 226 | 220
Days per Month | -1.85 (0.18) | -3.67 (0.22) | -3.63 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -1.82, 95% CI 2-sided [-2.29 to -1.36], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -1.78, 95% CI 2-sided [-2.25 to -1.31], Standard Error of Mean 0.24

5. Secondary Outcome: Mean Change From Baseline in Patient Global Impression of Severity (PGI-S) Rating
Description: The PGI-S scale is a participant-rated instrument that measures patients own global impression of their illness severity. The participant was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options were from 1 ("normal, not at all ill") to 7 ("extremely ill"). Mean is derived from the average of months 4 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 4 through Month 6
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months subcutaneous injection.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 443 | 226 | 219
units on a scale | -0.94 (0.07) | -1.22 (0.08) | -1.17 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p = .002, Mixed Models Analysis; LSMean Difference = -0.29, 95% CI 2-sided [-0.47 to -0.11], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p = .012, Mixed Models Analysis; LSMean Difference = -0.23, 95% CI 2-sided [-0.41 to -0.05], Standard Error of Mean 0.09

6. Secondary Outcome: Overall Mean Change From Baseline in Headache Hours
Description: Headache Hours is calculated as the total number of headache hours on which a headache occurred. Overall mean is derived from the average of months 1 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month and baseline MHD category.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Headache Hours per Month
Groups:
- Galcanezumab120mg: Participants received loading dose of 240mg galcanezumab followed by 120mg galcanezumab once a month for 5 months subcutaneously.
Arm/Group | Placebo | Galcanezumab120mg | Galcanezumab 240mg
Number analyzed (Participants) | 450 | 226 | 220
Headache Hours per Month | -10.89 (1.92) | -26.07 (2.41) | -24.44 (2.44)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -15.19, 95% CI 2-sided [-20.27 to -10.11], Standard Error of Mean 2.59
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -13.56, 95% CI 2-sided [-18.67 to -8.44], Standard Error of Mean 2.60

7. Secondary Outcome: Mean Change From Baseline in the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability.
  LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Galcanezumab120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months subcutaneous injection.
Arm/Group | Placebo | Galcanezumab120mg | Galcanezumab 240mg
Number analyzed (Participants) | 409 | 216 | 215
units on a scale | -12.02 (1.27) | -21.17 (1.58) | -20.24 (1.62)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -9.15, 95% CI 2-sided [-12.61 to -5.69], Standard Error of Mean 1.76
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -8.22, 95% CI 2-sided [-11.71 to -4.72], Standard Error of Mean 1.78

8. Secondary Outcome: Percentage of Participants Developing Anti-drug Antibodies (ADA) to Galcanezumab
Description: Treatment emergent (TE) ADA evaluable participant is considered to be TE ADA+ if the subject has at least one post-baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post-baseline result of ADA present with titer >= 1: 20.
Time Frame: Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug & had least one non-missing test result for ADA for each of the baseline period and the post-baseline period. As pre-specified in the analysis plan, outcome measures will not be reported for the ME2 arms/groups but only for the main global study arms/groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 443 | 222 | 214
percentage of participants | 0.45 | 8.56 | 5.14
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; TE ADA Positive; Test type: Superiority; p < .001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; TE ADA Positive; Test type: Superiority; p < .001, Fisher Exact

9. Secondary Outcome: Pharmacokinetics (PK): Serum Concentrations of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentrations of Galcanezumab.
Time Frame: Month 6
Population: All randomized participants who received at least one dose of study drug and had measurable serum concentrations.
  As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months subcutaneous injection.
Arm/Group | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 194 | 193
Nanogram per milliliter (ng/mL) | 17400 (8820) | 32200 (12600)

10. Secondary Outcome: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP).
Time Frame: Month 6
Population: All randomized participants who had received at least one dose of study drug and had measurable plasma concentration.
  As pre-specified in the analysis plan, outcome measures will not be reported for the Maximum Extended Enrollment (ME2) arms/groups but only for the main global study arms/groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months subcutaneously.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 29 | 187 | 185
ng/mL | 0.541 (1.11) | 3.93 (1.83) | 4.98 (1.60)

ADVERSE EVENTS:
Time Frame: Up to 10 Months
Description: There were 5 participants in Galcanezumab 120mg treatment phase, 1 participant in Galcanezumab 120mg post- treatment , 1 participant in Galcanezumab 120 mg treatment phase ME2 & 1 participant in Galcanezumab 120mg post-treatment ME2 arms who discontinued after receiving loading dose of 240mg, these participants were included in Galcanezumab 240mg Treatment, Post Treatment & equivalent ME2 arms for adverse event reporting.
  Per protocol, AE analysis was planned per treatment regimen received.
Groups:
- Placebo - Treatment Phase; Placebo - Treatment Phase ME2: Participants received placebo subcutaneously once a month for 6 months.
- Galcanezumab 120mg - Treatment Phase; Galcanezumab 120mg - Treatment Phase ME2: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months subcutaneously.
- Galcanezumab 240mg - Treatment Phase; Galcanezumab 240mg - Treatment Phase ME2: Participants received 240mg galcanezumab subcutaneously once a month for 6 months.
- Placebo - Post-treatment Phase; Galcanezumab 120mg - Post-treatment Phase; Galcanezumab 240mg - Post-treatment Phase; Placebo - Post-treatment Phase ME2; Galcanezumab 120mg - Post-treatment Phase ME2; Galcanezumab 240mg - Post-treatment Phase ME2: Participants didn't receive any intervention.
Arm/Group | Placebo - Treatment Phase | Galcanezumab 120mg - Treatment Phase | Galcanezumab 240mg - Treatment Phase | Placebo - Post-treatment Phase | Galcanezumab 120mg - Post-treatment Phase | Galcanezumab 240mg - Post-treatment Phase | Placebo - Treatment Phase ME2 | Galcanezumab 120mg - Treatment Phase ME2 | Galcanezumab 240mg - Treatment Phase ME2 | Placebo - Post-treatment Phase ME2 | Galcanezumab 120mg - Post-treatment Phase ME2 | Galcanezumab 240mg - Post-treatment Phase ME2
All-Cause Mortality (participants affected / at risk) | 0/461 | 0/226 | 0/228 | 0/410 | 0/212 | 0/208 | 0/30 | 0/14 | 0/20 | 0/25 | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 5/461 | 5/226 | 7/228 | 3/410 | 1/212 | 3/208 | 1/30 | 1/14 | 0/20 | 2/25 | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 150/461 | 78/226 | 87/228 | 40/410 | 16/212 | 13/208 | 10/30 | 9/14 | 9/20 | 3/25 | 6/14 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Treatment Phase (N=461) | Galcanezumab 120mg - Treatment Phase (N=226) | Galcanezumab 240mg - Treatment Phase (N=228) | Placebo - Post-treatment Phase (N=410) | Galcanezumab 120mg - Post-treatment Phase (N=212) | Galcanezumab 240mg - Post-treatment Phase (N=208) | Placebo - Treatment Phase ME2 (N=30) | Galcanezumab 120mg - Treatment Phase ME2 (N=14) | Galcanezumab 240mg - Treatment Phase ME2 (N=20) | Placebo - Post-treatment Phase ME2 (N=25) | Galcanezumab 120mg - Post-treatment Phase ME2 (N=14) | Galcanezumab 240mg - Post-treatment Phase ME2 (N=20)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/393 (0) | 1/192 (1) | 0/196 (0) | 0/349 (0) | 0/179 (0) | 0/181 (0) | 0/22 (0) | 0/13 (0) | 0/14 (0) | 0/18 (0) | 0/13 (0) | 0/14 (0) — All randomized female participants.
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/393 (0) | 0/192 (0) | 0/196 (0) | 0/349 (0) | 1/179 (1) | 0/181 (0) | 0/22 (0) | 0/13 (0) | 0/14 (0) | 0/18 (0) | 0/13 (0) | 0/14 (0) — All randomized female participants.
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Treatment Phase (N=461) | Galcanezumab 120mg - Treatment Phase (N=226) | Galcanezumab 240mg - Treatment Phase (N=228) | Placebo - Post-treatment Phase (N=410) | Galcanezumab 120mg - Post-treatment Phase (N=212) | Galcanezumab 240mg - Post-treatment Phase (N=208) | Placebo - Treatment Phase ME2 (N=30) | Galcanezumab 120mg - Treatment Phase ME2 (N=14) | Galcanezumab 240mg - Treatment Phase ME2 (N=20) | Placebo - Post-treatment Phase ME2 (N=25) | Galcanezumab 120mg - Post-treatment Phase ME2 (N=14) | Galcanezumab 240mg - Post-treatment Phase ME2 (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (15) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 39 (142) | 21 (100) | 20 (61) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 7 (17) | 18 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (12) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 14 (16) | 3 (4) | 9 (9) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 41 (49) | 19 (23) | 16 (21) | 18 (19) | 5 (5) | 4 (5) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (19) | 13 (14) | 12 (12) | 3 (4) | 4 (5) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0/393 (0) | 2/192 (2) | 1/196 (1) | 2/349 (2) | 0/179 (0) | 0/181 (0) | 0/22 (0) | 0/13 (0) | 1/14 (1) | 0/18 (0) | 0/13 (0) | 0/14 (0) — All randomized female participants.
Vulvovaginitis (Infections and infestations) | 1/393 (1) | 0/192 (0) | 0/196 (0) | 0/349 (0) | 0/179 (0) | 0/181 (0) | 0/22 (0) | 0/13 (0) | 1/14 (1) | 0/18 (0) | 0/13 (0) | 0/14 (0) — All randomized female participants.
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (24) | 2 (2) | 5 (5) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (12) | 8 (10) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (9) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/393 (0) | 0/192 (0) | 0/196 (0) | 0/349 (0) | 1/179 (1) | 0/181 (0) | 0/22 (0) | 1/13 (2) | 0/14 (0) | 0/18 (0) | 0/13 (0) | 0/14 (0) — All randomized female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02614196/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT02614196/SAP_001.pdf